CLINICAL TRIAL: NCT04293146
Title: Pre- Versus Sub-pectoral Implant-based Breast Reconstruction After Skin-sparing Mastectomy or Nipple-sparing Mastectomy (OPBC-02/ PREPEC): a Pragmatic, Multicenter, Randomized, Superiority Trial
Brief Title: Pre- Versus Sub-pectoral Implant-based Breast Reconstruction After Skin-sparing Mastectomy or Nipple-sparing Mastectomy OPBC-02PREPEC
Acronym: OPBC-02PREPEC
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Basel, Switzerland (Other)
Collaborators: Swiss National Science Foundation (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: 2020-00256; ch18Weber4
Record Dates: First submitted 2020-02-21; First posted 2020-03-03 (Actual); Last update posted 2024-12-13 (Actual); Status verified 2024-12

CONDITIONS: Breast Reconstruction; Implant-Based Breast Reconstruction (IBBR)
Keywords: skin-sparing mastectomy (SSM); nipple-sparing mastectomy (NSM); immediate breast reconstruction; pre-pectoral breast implant; sub-pectoral breast implant

STUDY DESIGN:
Intervention Model Description: The study will objectively assess the results and complication of two surgical techniques and thus provide evidence to assess whether there are differences between these techniques.
Who Masked: Outcomes Assessor
Masking Description: blinded outcome assessment for aesthetic results
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- pre-pectoral IBBR (Active Comparator)
  Interventions: Procedure: pre-pectoral IBBR
- sub-pectoral IBBR (Active Comparator)
  Interventions: Procedure: sub-pectoral IBBR

INTERVENTIONS:
Procedure: pre-pectoral IBBR — The breast is reconstructed by positioning a breast implant above (pre-pectoral) the pectoralis major muscle.
  Arms: pre-pectoral IBBR
Procedure: sub-pectoral IBBR — The breast is reconstructed by positioning a breast implant below (sub-pectoral) the pectoralis major muscle.
  Arms: sub-pectoral IBBR

SUMMARY:
This trial is to investigate whether pre-pectoral Implant-Based Breast Reconstruction (IBBR) provides better Quality of Life (QoL) with respect to long-term (24 months) physical well-being (chest) compared to sub-pectoral IBBR for patients undergoing skin-sparing mastectomy or nipple-sparing mastectomy for prevention or treatment of breast cancer.

DETAILED DESCRIPTION:
This trial is to investigate whether pre-pectoral Implant-Based Breast Reconstruction (IBBR) provides better Quality of Life (QoL) with respect to long-term (24 months) physical well-being (chest) compared to sub-pectoral IBBR for patients undergoing skin-sparing mastectomy or nipple-sparing mastectomy for prevention or treatment of breast cancer.The aim is to adhere to standard of care as much as possible to follow the pragmatic trial design to generate data that are applicable to today's practice. Therefore, surgeons are allowed to use their preferred Acellular Dermal Matrix (ADM), synthetic meshes, expanders and implants, thereby offering practitioners considerable leeway in deciding how to perform the procedure. For the same reason, both the one- and two-staged IBBR approaches are allowed when studying pre- versus sub-pectoral IBBR.

ELIGIBILITY:
Inclusion Criteria:

* Written informed consent according to ICH/GCP regulations prior to any trial specific procedures
* Patients undergoing NSM or SSM and IBBR in the therapeutic or risk-reducing Setting
* Ability to complete the Quality of Life questionnaires

Exclusion Criteria:

* No indication for IBBR according to clinical judgment of the treating surgeon
* Skin flaps inadequate for pre-pectoral IBBR.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 382 (Actual)
Dates: Start 2020-07-28 (Actual); Primary Completion 2025-05 (Estimated); Study Completion 2033-02 (Estimated)

PRIMARY OUTCOMES:
Change in BREAST-Q scale | within 24 months after mastectomy (screening, day 10, and months 1, 6, 12 and 24)
  compare the Quality of Life (QoL) with respect to long-term physical well-being (chest) after pre-pectoral or sub-pectoral IBBR. The BREAST-Q module specific to breast reconstruction version 2.0 consists of 13 independent scales covering health-related QoL domains and satisfaction domains. Each scale is scored to generate a numerical score on a scale from 0 (worst) to 100 (best).
Change in EQ-5D-5L questionnaire | within 24 months after mastectomy (screening, day 10, and months 1, 6, 12 and 24)
  The 5-level version of the EQ-5D (EQ-5D-5L) consists of the EQ-5D descriptive system that comprises five dimensions: mobility, self-care, usual activities, pain/discomfort and anxiety/Depression (5 answer levels each: no problems, slight problems, moderate problems, severe problems and extreme problems), resulting in a 1-digit number that expresses the level for that dimension. The digits for each dimension are combined into a 5-digit number that describes the patient's health state and is subsequently converted into a preference-based quality of life weight (utility) using an algorithm derived from population-based studies. In addition, patients are asked to rate their health on a vertical visual analogue scale (EQ VAS), where the anchors are labelled with 'The best health you can imagine' and 'The worst health you can imagine'.

SECONDARY OUTCOMES:
loss of expander or implant | within 24 months of undergoing mastectomy and immediate reconstruction
  compare the safety of pre-pectoral and sub-pectoral IBBR, in terms of loss of expander or implant. Loss of expander or implant is defined as an unplanned surgical removal of expander/implant with or without immediate replacement.
surgical complications | within 24 months of undergoing mastectomy and immediate reconstruction
  compare the safety of pre-pectoral and sub-pectoral IBBR, in terms of surgical complications. The complications include: Wound dehiscence, Haematoma, Seroma, Implant/expander exposure/Extrusion, Implant/Expander rotation/malpositioning, Infection, Mastectomy skin flap necrosis, Capsular contraction, Lymphedema
thromboembolic events | within 24 months of undergoing mastectomy and immediate reconstruction
  compare the safety of pre-pectoral and sub-pectoral IBBR, in terms of thromboembolic events according to Common Terminology Criteria for Adverse Events (CTCAE) v5.0
patient satisfaction | over 24 months since mastectomy
  compare patient satisfaction after pre-pectoral or sub-pectoral IBBR
animation deformity | before and 24 months after the mastectomy
  compare animation deformity after pre-pectoral or sub-pectoral IBBR by using pictures from before and 24 months after the mastectomy
capsular contracture | before and 24 months after the mastectomy
  compare capsular contracture after pre-pectoral or sub-pectoral IBBR by using pictures from before and 24 months after the mastectomy
aesthetic results | before and 24 months after the mastectomy
  compare aesthetic results after pre-pectoral or sub-pectoral IBBR assessed by photographs of the breast taken in a standardized way. They will be evaluated by an experienced investigator who is blinded for group assignment. The blinded outcome assessment team will be trained to enter data for the two most widely used semi-automatic software for objective aesthetic evaluation, the 'Breast Cancer Conservative Treatment cosmetic results' (BCCT.core)
Recurrence-free survival (RFS) | until 10 years after mastectomy and IBBR.
  RFS is defined as the time from randomization until the first documentation of any of the following events: local-regional occurrence or recurrence of invasive disease or ductal carcinoma in situ (DCIS), distant breast cancer metastasis, or death from any cause.
aesthetic results evaluated by patients | at baseline and after 24 months
  evaluated by patients using a four point scale: excellent, good, regular, bad.
total number of operative procedures | until 24 months after mastectomy
  assess the burden on patients by total number of operative procedures
length of hospital stay (index hospitalization and overall) | until 24 months after randomization
  length of hospital stay (index hospitalization and overall) following randomization until discharge and the cumulative number of days the patient was hospitalized
total number of outpatient visits at the trial site and the emergency department | from admission for mastectomy until 24 months after randomization
  assess the burden on patients by total number of outpatient visits at the trial site and the emergency department
aesthetic results evaluated by local physicians | at baseline and after 24 months
  evaluated by local physicians using a four point scale: excellent, good, regular, bad.

CONTACTS AND LOCATIONS:
Overall Officials: Walter Weber, Prof. Dr. med, Principal Investigator — Division of Breast Surgery, University Hospital Basel
Locations (22):
- Brigham and Women's Hospital Harvard Medical School, Boston, Massachusetts, United States
- Austria (2):
  - Universitätsklinik für Frauenheilkunde und Geburtshilfe, Salzburg
  - Medizinische Universität Wien, Vienna
- Germany (4):
  - Evangelisches Krankenhaus BETHESDA zu Duisburg GmbH, Klinik für Frauenheilkunde, Geburtshilfe, Gynäkologische Onkologie & Senologie, Duisburg
  - KEM | Evang. Kliniken Essen-Mitte, Essen
  - Universitätsklinikum Heidelberg, Heidelberg
  - Landesfrauenklinik, Senologie und Brustzentrum, Wuppertal
- National Institute of Oncology, Budapest, Hungary
- Italy (2):
  - Universitario "Agostino Gemelli" di Roma, Unità Operativa di Chirurgia Senologica, Roma
  - Ospedale Santa Chiara, Breast Surgical Oncology/Oncoplastic Surgery. Breast Center, Trento
- Sweden (3):
  - Capio S:t Görans Hospital, Stockholm
  - Södersjukhuset, Stockholm
  - Karolinska University Hospital, Stockholm
- Switzerland (9):
  - Klinik Hirslanden Brustzentrum Aarau, Aarau
  - Kantonsspital Aarau AG, Aarau
  - University Hospital Basel, Division of Breast Surgery, Basel
  - Universitätsklinik für Plastische- und Handchirurgie, Inselspital, Bern
  - Lindenhof Bern, Bern
  - Kantonsspital Frauenfeld, Frauenfeld
  - Gesundheitszentrum Fricktal, Rheinfelden
  - Ospedale Regionale di Lugano, Viganello
  - Brust-Zentrum Zürich, Zurich

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Kappos EA, Schulz A, Regan MM, Moffa G, Harder Y, Ribi K, Potter S, Pusic AL, Fehr MK, Hemkens LG, Holzbach T, Farhadi J, Simonson C, Knauer M, Verstappen R, Bucher HC, Zwahlen D, Zimmermann F, Schwenkglenks M, Mucklow R, Shaw J, Bjelic-Radisic V, Chiorescu A, Chun YS, Farah S, Xiaosong C, Nigard L, Kuemmel S, Reitsamer R, Hauschild M, Fulco I, Tausch C, Fischer T, Sarlos D, Constantinescu MA, Lupatsch JE, Fitzal F, Heil J, Matrai Z, de Boniface J, Kurzeder C, Haug M, Weber WP. Prepectoral versus subpectoral implant-based breast reconstruction after skin-sparing mastectomy or nipple-sparing mastectomy (OPBC-02/ PREPEC): a pragmatic, multicentre, randomised, superiority trial. BMJ Open. 2021 Sep 2;11(9):e045239. doi: 10.1136/bmjopen-2020-045239. PMID 34475143